CLINICAL TRIAL: NCT07058753
Title: An Intense Course of Prehabilitation in Ovarian Cancer Patients During Neoadjuvant Treatment Awaiting for Interval Debulking Surgery. PREHONED - a Prospective, Randomized, Multicentre Clinical Study.
Brief Title: Prehabilitation in Ovarian Cancer Patients During Chemiotherapy Before Cytoreductive Surgery.
Acronym: PREHONED
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Marcin Zębalski, MD, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREH/2025-2-1; PREH/2025-2-1 (Registry Identifier: Marcin Adam Zebalski)
Record Dates: First submitted 2025-06-23; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; prehabilitation; interval debulking surgery; neoadjuvant chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention group consists of patients undergoing prehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intense course of prehabilitation (Experimental): Patients undergoing intense prehabilitation program
  Interventions: Procedure: Prehabilitation. An intensive prehabilitation for NACT patients
- Standard preoperative care (No Intervention): Patients with standard preoperative care

INTERVENTIONS:
Procedure: Prehabilitation. An intensive prehabilitation for NACT patients — Patients referred to NACT (neoadjuvant chemotheraphy) for advanced ovarian cancer will undergo an intensive course of prehabilitation including physical exercise, a high-protein diet, protein and vitamin supplementation, optimization of laboratory test results, and psychological support will be provided.
  Arms: Intense course of prehabilitation

SUMMARY:
Prehabilitation includes care for patients preparing for surgery. This is a modern approach aimed at increasing the patient's functional capacity before surgery and improving postoperative results. Prehabilitation includes preoperative physical activity, nutritional intervention, psychological support, cessation of stimulants and optimization of laboratory test results.

Many studies have shown a positive effect of prehabilitation on postoperative results, mainly reducing the number of postoperative complications and shortening the hospitalization time.

The assumed time of prehabilitation is 2-6 weeks, but in the case of oncology patients, the procedure should not be delayed only for the sake of prehabilitation.

Our study includes oncology patients with ovarian cancer who are referred for neoadjuvant chemotherapy before interval cytoreductive surgery. The assumption of the study is an intensive course of prehabilitation during neoadjuvant treatment, which should provide significantly better postoperative results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed ovarian cancer
* No possibility of performing primary debulking surgery (Fagotti score > 8 points). Referral patient for neoadjuvant chemotherapy
* Consent to participate in the study
* Age over 18 years

Exclusion Criteria:

* Performing primary debulking surgery
* Lack of consent to participate in the study
* Aletti score < 4 points in interval debulking surgery
* Severe neurological/psychiatric disorders that make contact with the patient difficult

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of postoperative complications | from surgery for the next 30 days
  Analysis of the incidence of complications, including assessment according to the Clavien-Dindo classification. Analysis of complications will include the incidence of intensive care units hospitalization, frequency of reoperation, dehiscence of intestinal anastomosis, wound dehiscence with eventeration, need for blood transfusion and readmission within 30 days
Length of hospital stay | from surgery to hospital discharge (assessed up to 14 days)
  The analysis will include the length of hospitalization after surgery.
Time to start adjuvant chemotherapy | from discharge from hospital for the next 2 months
  Comparison of time from hospital discharge to start of adjuvant chemotherapy

SECONDARY OUTCOMES:
Progression-free survival | From the time of the operation for the next 3 and 5 years
  Comparison of progression-free survival in both groups at 3 and 5 years of follow-up.
Overall survival | From the time of the operation for the next 3 and 5 years
  Comparison of overall survival in both groups at 3 and 5 years of follow-up

OTHER OUTCOMES:
Quality of life assessment | From study enrollment to surgery (up to 4 months)
  Measuring changes in quality of life during the prehabilitation program. The assessment of quality of life will be performed using the standardized EORTC Quality of Life QLQ-C30 questionnaire. The EORTC QLQ-C30 assesses quality of life in five functional domains (physical, role, cognitive, emotional, and social), three symptom domains (fatigue, pain, nausea and vomiting), a global health status domain (GHS/QoL), and five single-item domains (dyspnoea, insomnia, loss of appetite, constipation and diarrhea, and financial problems due to illness) The higher the score in the functional domains and in the global health status domain, the better the patient's quality of life, while the higher the score in the symptom domain, the worse the quality of life due to the severity of disease-related symptoms.
Depression and anxiety assessment | from study enrollment to surgery (up to 4 months)
  Measuring changes in depression and anxiety during the prehabilitation program. The assessment of depression and anxiety will be performed using the HADS questionnaire. The HADS is a self-report questionnaire, and it consists of 2 subscales designed to identify and quantify anxiety and depression in patients, especially in oncological patients whereas a score of 8 points indicates mild anxiety or depression and the higher the score, the greater the severity of anxiety and depressive disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Nowosielski, MD, PhD, Study Chair — Department of Gynecology, Obstetrics and Gynecological Oncology, University Clinical Center of the Medical University of Silesia; Marcin A Zębalski, MD, Principal Investigator — Department of Gynecology, Obstetrics and Gynecological Oncology, University Clinical Center of the Medical University of Silesia
Locations (1):
- Department of Gynecology, Obstetrics and Gynecological Oncology, University Clinical Center of the Medical University of Silesia, Katowice, Poland

IPD SHARING:
Plan to Share IPD: Undecided